CLINICAL TRIAL: NCT00337584
Title: A Pre-Operative Screening Questionnaire (AMS-Q) for Ambulatory Orthopedic Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 24003
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Ambulatory Surgery
Keywords: out patient surgery; quality improvement

INTERVENTIONS:
Procedure: Pre-surgical screening

SUMMARY:
We are studying whether providing patients undergoing day surgery the opportunity to have their medical history reviewed by an hospital internist before surgery leads to better results after surgery. These doctors are internal medicine specialists who are experienced in assessing patients going to surgery, making sure they are "fine-tuned" before their operation. We believe this will ensure the safest and best surgical outcomes. The study involves the patient filling out a 3 page questionnaire for review by the internist prior to surgery. Additionally, patients will receive a follow-up phone call one week after surgery asking about the experience at the hospital and a questionnaire in the mail three months later to see if the patient had any medical problems after leaving the hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients having ambulatory surgery performed by one of our participating surgeons during the study period.

Exclusion Criteria:

* Patients who speak neither English nor Spanish.
* Patients who have had any surgery in the previous 6 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-12; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Mandl, MD MPH, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States